CLINICAL TRIAL: NCT03755869
Title: An Open, Single-arm, Multi-center Study of Anlotinib in Non-squamous NSCLC Patients Who Failed First-Line Chemotherapy
Brief Title: Study of Anlotinib in Non-squamous NSCLC Patients Who Failed First-Line（ALTER-L020）
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tang-Du Hospital (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2018LSK-073
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2019-04

CONDITIONS: Non-squamous NSCLC
Keywords: Non-squamous NSCLC; Anlotinib
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib ( 12mg, QD, PO, d1-14, 21 days per cycle), take once when limosis in the morning. If patients cannot suffer from AEs, they can get declined dosage.
  Other Names: AL3818

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor celltebiz related kinase -c-Kit kinase. In the phase III study, Patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib (12mg, po. qd. on day 1to14 of a 21-day cycle) or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months.

DETAILED DESCRIPTION:
It is an open, single-arm, multi-center clinical trial conducted in China, and plan to Recruiting103 patients who were progressed after first line systemic therapy and refused/can't tolerate chemotherapy. Patents receive 12mg anlotinib orally daily on day 1to 14 of a 21-day cycle until progression of disease, assess safety and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Age：18~75 years;
* Subjects with histologically or cytologically confirmed locally advanced and/or advanced NSCLC
* at least two systematic chemotherapy with upwards of 1-line treatments or cannot suffer
* The negative patients in EGFR&ALK can participate or who positive in EGFR&ALK, have or have not drug tolerance after the treatment with relative targeted drugs
* Subjects with at least one measurable lesion as defined by RECIST (version 1.1)
* Expected Survival Time: Over 3 months
* ECOG PS：0-1,
* main organs function is normal
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it

Exclusion Criteria:

* 1.Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
* lung squamous carcinoma
* Other active malignancies requiring treatment
* History of malignancy
* Have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* Abnormal coagulation (INR>1.5 or PT>ULN+4s or APTT >1.5 ULN); Patients with any physical signs of bleeding diathesis or receiving thrombolysis and anticoagulation
* take major surgical treatments or have serious trauma before grouping, or the impact of surgery or trauma has been eliminated for less than 14 days.
* Patients with active or unable to control serious infections;
* Patients with Grade II or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc male ≥ 450 ms, female ≥ 470 ms) ; Patients with grade III to IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) <50% (NYHA Classification)
* Patients with non-healing wounds or fractures
* with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus).
* get arterial/venous thrombosis within 12 months, such as cerebrovascular accidents (including temporary ischemic stoke), deevenous thrombosis, and pulmonary embolism
* plan to take systemic anti-tumor therapy within 4 weeks before grouping or during the medicine-taking period of this research, including Cytotoxic Therapy, Signal Transduction Inhibitor, and Immunotherapy
* Patients with cirrhosis, decompensated liver disease, or active hepatitis Have suffered from hemorrhagic disease or coagulation dysfunction
* diagnosed with disease which will severely endanger the security of patients or influence the completion of this research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Duration of Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1 | Baseline until PD or death, whichever occurs first (up to approximately 24 months)
  Progress free survival (PFS)

SECONDARY OUTCOMES:
Duration of Overall Survival (OS) as Assessed by the Investigator Using RECIST v1.1 | Baseline until death from any cause (up to approximately 24 months)
  Overall Survival (OS)
Disease Control Rate (DCR)as Assessed by the Investigator Using RECIST v1.1 | First occurrence of PR or CR until PD or death, whichever occurs first (up to 24 months)
  Disease Control Rate (DCR)
Objective Response Rate (ORR) as Assessed by the Investigator Using RECIST v1.1 | Baseline until partial response (PR) or complete response (CR), whichever occurs first (up to 24 months)
  Objective Response Rate (ORR)
Percentage of Participants with Adverse Events | Baseline until up to 21 days after end of treatment
  Percentage of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: enxiao li, professor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Shaanxi Provincial Cancer Hospital, Xian, Shanxi, China

IPD SHARING:
Plan to Share IPD: No